CLINICAL TRIAL: NCT06554613
Title: An Open-label, Two-arm, Multicenter, Phase II Randomized Controlled Trial Assessing the Impact of Olanzapine on the Efficacy of First-line Immunotherapy in Patients With Advanced EGFR Mutation-negative Non-small Cell Lung Cancer (NSCLC).
Brief Title: Olanzapine Impact on First-line Immunotherapy for Advanced EGFR-negative NSCLC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2024-6804
Record Dates: First submitted 2024-07-02; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-06

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Olanzapine; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Olanzapine in Combination with Immune Checkpoint Inhibitors Treatment Group (Experimental): Receiving first-line treatment with a PD-1/PD-L1 inhibitor as a single agent or in combination with chemotherapy (according to the instructions manual)，Medication is administered on the first day of each cycle, with one cycle every 3 weeks. A continuous 21-day treatment constitutes one treatment cycle.Then receive olanzapine orally at a dose of 5mg once daily (qd), with continuous administration for 6-8 weeks.
  Interventions: Drug: Olanzapine; Drug: Nivolumab
- Group Without Olanzapine (Active Comparator): Receiving first-line treatment with a PD-1/PD-L1 inhibitor as a single agent or in combination with chemotherapy (according to the instructions manual)，Medication is administered on the first day of each cycle, with one cycle every 3 weeks. A continuous 21-day treatment constitutes one treatment cycle..
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Olanzapine — Olanzapine 5mg qd (once daily), q3w(every 3 weeks), oral therapy，Administered continuously for 6-8 weeks.
  Other Names: Zyprexa
  Arms: Olanzapine in Combination with Immune Checkpoint Inhibitors Treatment Group
Drug: Nivolumab — Nivolumab，Infused intravenously once every 3 weeks at a dose of 2mg/kg, with a continuous 21-day treatment period constituting one treatment cycle.
  Other Names: Opdivo

SUMMARY:
Clinical Trial

The objective of this clinical trial is to determine whether antidepressant medications, such as olanzapine, in combination with immune checkpoint inhibitors are more effective than the use of immune checkpoint inhibitors alone. The main questions it aims to answer are:

Is the combination therapy of antidepressant medication with immune checkpoint inhibitors more efficacious than the therapy with immune checkpoint inhibitors alone? What medical issues might participants encounter when treated with the combination of antidepressant medication and immune checkpoint inhibitors?

Participants will:

Take olanzapine in combination with immune checkpoint inhibitors or immune checkpoint inhibitors alone for 2 months.

Visit the clinic for check-ups and tests every two weeks, and have follow-up visits every six weeks after the treatment ends.

Keep a record of their symptoms and disease progression.

DETAILED DESCRIPTION:
An Open-label, Two-arm, Multicenter, Phase II Randomized Controlled Study on the Impact of Olanzapine on the Efficacy of First-line Immunotherapy in Patients with Advanced EGFR Mutation-negative Non-small Cell Lung Cancer (NSCLC).

Primary Research Objective:

To evaluate the objective response rate (ORR) in patients with advanced EGFR mutation-negative NSCLC treated with first-line PD-1/PD-L1 inhibitors combined with olanzapine.

Secondary Research Objectives:

To evaluate the interval of progression-free survival (iPFS) in patients with advanced EGFR mutation-negative NSCLC treated with first-line PD-1/PD-L1 inhibitors combined with olanzapine.

To evaluate other antitumor efficacy indicators in patients with advanced EGFR mutation-negative NSCLC treated with first-line PD-1/PD-L1 inhibitors combined with olanzapine: progression-free survival (PFS), duration of response (DoR), and disease control rate (DCR).

To assess the safety (Safety) and the improvement of quality of life (QoL) in patients with advanced EGFR mutation-negative NSCLC treated with first-line PD-1/PD-L1 inhibitors combined with olanzapine.

To explore the impact of antipsychotic medication on the immune response to first-line immunotherapy in advanced NSCLC.

Study Design:

This study is an open-label, two-arm, multicenter, phase II randomized controlled study designed to evaluate and observe the impact of olanzapine on the efficacy of first-line immunotherapy in patients with advanced EGFR mutation-negative NSCLC. Eligible participants who meet all inclusion criteria and do not meet any exclusion criteria will receive first-line treatment with PD-1/PD-L1 monoclonal antibodies alone or in combination with chemotherapy (according to the instructions for use).

Study Subjects:

Ages 18 years and above (including 18) and up to 75 years (including 75); histologically or cytologically confirmed EGFR mutation-negative NSCLC; intended to receive first-line treatment with PD-1/PD-L1 inhibitors alone or in combination with chemotherapy.

Inclusion Criteria:

Participants voluntarily join this study and sign an informed consent form, with good compliance and cooperation with follow-up.

Age is 18 years and above (including 18) and up to 75 years (including 75). ECOG score: 0-2 points. Expected survival is no less than 3 months. Staged as Stage IV according to the TNM system. Confirmed to have NSCLC with EGFR mutation-negative by histology or cytology. Has not received systemic antitumor treatment, and is intended to receive first-line treatment with PD-1/PD-L1 inhibitors alone or in combination with chemotherapy.

Normal major organ function, that is, meeting the following criteria: (1) Hematological examination criteria must be met: Hb≥90 g/L; ANC≥1.5×10^9/L; PLT≥80×10^9/L. (2) Biochemical examination must meet the following criteria: TBIL<1.5ULN; ALT and AST<2.5ULN; serum Cr≤1.25ULN or endogenous creatinine clearance > 45 ml/min (Cockcroft-Gault formula).

Women of childbearing age must have taken reliable contraceptive measures and have undergone a pregnancy test (serum or urine) within 7 days before enrollment, with a negative result, and are willing to use appropriate methods of contraception during the trial period and for 8 weeks after the last administration of the trial medication. For men, they must agree to use appropriate methods of contraception during the trial period and for 8 weeks after the last administration of the trial medication or have undergone surgical sterilization.

Data Analysis/Statistical Methods:

Common Analysis This study will summarize the data using corresponding descriptive statistics according to the type of data, that is, for quantitative data, mean (Mean), standard deviation (SD), median (Median), minimum value (Minimum), and maximum value (Maximum) will be used, and for count data and grade data, frequency and percentage will be used, and time-event data will be estimated by the Kaplan-Meier method for the median time and the overall 95% confidence interval.

Efficacy Analysis The primary efficacy endpoint, the objective response rate (ORR) based on the investigator's assessment, will be compared between groups using the Fisher's exact probability test and the two-sided 95% confidence interval will be listed.

The secondary efficacy indicators, including the interval of progression-free survival (iPFS), progression-free survival (PFS), duration of response (DoR), and disease control rate (DCR), will be estimated using the Kaplan-Meier method for the median time and the median event and the two-sided 95% confidence interval will be listed, and the hazard ratio and its 95% confidence interval will be estimated. The disease control rate (DCR = CR + PR + SD) will be compared between groups using Fisher's exact probability test and the two-sided 95% confidence interval will be listed. Quality of life score statistical tests will use ANOVA or two-sided t-tests, and a P-value less than or equal to 0.05 will be considered statistically significant. Comparisons of changes before and after within groups will be made using paired t-tests.

Safety Analysis Safety analysis will mainly summarize descriptive statistics. Statistics will be summarized for adverse events (AEs) and treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), and laboratory data, vital signs, etc. At the same time, statistical summaries will be made for the exposure to the study drug (including treatment cycles, total dose received, and dose intensity). The above data will be analyzed and summarized according to the current clinical trial reporting standards. Including: summary of adverse events (all causes and related to treatment); incidence and severity of adverse events (all causes and related to treatment); analysis of adverse events related to the drug; analysis of the outcome of adverse events; analysis of serious adverse events.

Sample Size Estimation:

This study is an open-label, two-arm, multicenter, phase II randomized controlled study. The primary research objective is to evaluate the objective response rate (ORR) in patients with advanced EGFR mutation-negative NSCLC treated with first-line PD-1/PD-L1 inhibitors combined with olanzapine. The study endpoint is the objective response rate (ORR) of the patients. Referring to historical literature, the ORR of first-line chemotherapy combined with immunotherapy in advanced NSCLC patients is about 50%, and it is expected that the combination with olanzapine can increase the ORR by 15%. After the first subject is enrolled, the longest observation period is 24 months, with α being two-sided 0.05, and the power being 90%, the study plans to enroll 156 subjects, with 78 in the experimental group and 78 in the control group, calculated with a 10% loss to follow-up rate.

ELIGIBILITY:
Inclusion Criteria:

1. Participants voluntarily enroll in this study and sign an informed consent form, with good compliance and cooperation with follow-up.
2. Age is over 18 years old (including 18 years old) and under 75 years old (including 75 years old).
3. ECOG score: 0-2 points.
4. Expected survival is no less than 3 months.
5. Staged as Stage IV according to the TNM system.
6. Histologically or cytologically confirmed EGFR mutation-negative non-small cell lung cancer.
7. Has not received systemic antitumor treatment, and is intended to receive monotherapy or combined chemotherapy with a PD-1/PD-L1 inhibitor as first-line treatment.
8. Normal major organ function, that is, meeting the following criteria: (1) Hematological examination criteria must be met: Hb≥90 g/L; ANC≥1.5×10^9/L; PLT≥80×10^9/L. (2) Biochemical examination must meet the following criteria: TBIL<1.5×ULN; ALT and AST<2.5×ULN; serum Cr≤1.25×ULN or endogenous creatinine clearance > 45 ml/min (Cockcroft-Gault formula).
9. Women of childbearing age must have taken reliable contraceptive measures and have undergone a pregnancy test (serum or urine) within 7 days before enrollment, with a negative result, and are willing to use appropriate methods of contraception during the trial period and for 8 weeks after the last administration of the trial medication. For men, they must agree to use appropriate methods of contraception during the trial period and for 8 weeks after the last administration of the trial medication or have undergone surgical sterilization.

Exclusion Criteria:

1. Have received any of the following treatments:

   1. Previously used any EGFR tyrosine kinase inhibitors;
   2. Previously received any chemotherapy for lung cancer;
   3. Previously received any radiotherapy for lung cancer (except palliative radiotherapy for bone metastases);
   4. Within 4 weeks prior to the first administration of the study drug, the subject had undergone major surgery;
   5. Within 7 days prior to the first administration of the study drug, used strong inhibitors or inducers of CYP3A4.
2. Subjects with concurrent other malignant tumors, except for basal cell carcinoma of the skin and in situ cancer.
3. Subjects with uncontrollable malignant pleural effusion and pericardial effusion.
4. Subjects allergic to contrast agents for CT and MRI or any subjects who cannot tolerate MRI examination.
5. As judged by the investigator, any serious or poorly controlled systemic diseases, such as uncontrolled hypertension, active bleeding diathesis, or active infection.
6. Clinically severe gastrointestinal functional abnormalities that may affect the intake, transport, or absorption of the drug, such as the inability to take oral medication, uncontrollable nausea or vomiting, history of extensive gastrointestinal resection, unresolved recurrent diarrhea, atrophic gastritis, gastric diseases requiring long-term use of proton pump inhibitors, Crohn's disease, ulcerative colitis, etc.
7. Hepatic encephalopathy, hepatorenal syndrome, or liver cirrhosis.
8. Meet any of the following cardiac examination results:

   1. The average of the corrected QT interval (QTcF) obtained from three ECG examinations at rest is > 470 msec;
   2. Resting ECG suggests conduction or ECG morphological abnormalities (such as complete left bundle branch block, third-degree atrioventricular block, second-degree atrioventricular block, and PR interval > 250 msec, etc.);
   3. There are any factors that increase the risk of QTc prolongation or arrhythmic events, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or any concurrent medication of unexplained sudden death in direct relatives under the age of 40 or prolonged QT interval;
   4. Left ventricular ejection fraction (LVEF) < 50%.
9. Insufficient bone marrow reserve or organ function, reaching any of the following laboratory limits:

   1. Absolute neutrophil count <1.5×10^9/L;
   2. Platelet count <100×10^9/L;
   3. Hemoglobin <90 g/L (<9 g/dL);
   4. If there is no definite liver metastasis, alanine aminotransferase > 3 times the upper limit of normal (ULN); if there is liver metastasis, alanine aminotransferase > 5×ULN;
   5. If there is no definite liver metastasis, aspartate aminotransferase >3×ULN; if there is liver metastasis, aspartate aminotransferase > 5×ULN;
   6. If there is no definite liver metastasis, total bilirubin > 1.5×ULN; or with Gilbert's syndrome (unconjugated hyperbilirubinemia) or liver metastasis, total bilirubin > 3×ULN;
   7. Creatinine > 1.5×ULN and creatinine clearance <50 mL/min (calculated by the Cockcroft-Gault formula); creatinine clearance is only required if creatinine > 1.5×ULN;
   8. Serum albumin (ALB) <28 g/L.
10. Active fungal, bacterial, and/or viral infections requiring systemic treatment.
11. Female subjects who are pregnant, breastfeeding, or planning to become pregnant during the study period.
12. History of interstitial lung disease, drug-induced interstitial lung disease, history of radiation pneumonitis requiring steroid treatment, or any evidence of clinically active interstitial lung disease.
13. Subjects who, in the judgment of the investigator, may have poor compliance with the procedures and requirements of the study, such as subjects with a clear history of neurological or mental disorders, currently suffering from mental disorders, etc.
14. Subjects whom the investigator judges to have any condition that endangers the safety of the subject or interferes with the evaluation of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
The Overall Survival（OS） | 24 months
  The Overall Survival（OS），From the time of a patient's diagnosis or the commencement of treatment, to the time of the patient's death.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Chuyang, Director, Study Director — Nanchang University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang M, Herbst RS, Boshoff C. Toward personalized treatment approaches for non-small-cell lung cancer. Nat Med. 2021 Aug;27(8):1345-1356. doi: 10.1038/s41591-021-01450-2. Epub 2021 Aug 12. PMID 34385702
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338